CLINICAL TRIAL: NCT03001934
Title: Super Chinese Nephrotic Syndrome Registration System (SUCCESS)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: SUCCESS
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic syndrome; Treatment response; Renal function
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The serum, urine, DNA and renal tissue will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nephrotic syndrome patients: Patients diagnosis as nephrotic syndrome (NS)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Registration of all NS patients in the First Affiliated Hospital of Sun Yat-sen University and other hospitals which have signed the contract in China.

SUMMARY:
The investigators are registering all nephrotic syndrome (NS) patients regardless of the primary causes and developing a NS database in China. Patients will be followed-up and both baseline and follow-up information will be recorded in the registration system. The treatment response, longitudinal changes of renal function, renal survival, patient survival, infection events and acute kidney injury etc, will be analyzed using the NS database.

DETAILED DESCRIPTION:
The investigators are registering all NS patients regardless of the primary causes in China. Patients' demographic characteristics (including age, gender, height, weight, BMI, smoking, drinking, and education), clinical characteristics (including systolic blood pressure, diastolic blood pressure, primary cause of NS, and lab measurements of serum, urine), pathological characteristics, treatment and treatment response, complications and outcomes. Patients will be followed up, the demographic, clinical characteristics, treatment, lab tests of blood and urine and complications of patients will be collected and recorded at each visit. The investigators also record the outcome at each visit, such as treatment response, longitudinal changes of renal function, hospitalization, occurrence of infection or cardiovascular events etc. The outcomes will be analyzed using the NS database.

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic syndrome patients regardless of the primary causes

Exclusion Criteria:

* No

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nephrotic syndrome patients
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-04; Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The patient survival in NS patients | 10 years

SECONDARY OUTCOMES:
Renal survival in NS patients | 10 years
  Renal survival including end stage renal disease, dialysis, renal transplantation
Longitudinal changes of renal function of NS patients | 10 years
Treatment response of NS patients | 10 years
Infection rate of NS patients | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes